CLINICAL TRIAL: NCT03877406
Title: Decrease in Body Fat and Increase in Ketone Body After 6-month Treatment of Empagliflozin in Korean Patients With Type 2 Diabetes
Brief Title: Effect of Empagliflozin on Body Composition and Ketones
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Division Chief of Endocrinology and Metabolism, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-1507/307-007
Record Dates: First submitted 2018-10-23; First posted 2019-03-15 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus; Fat; Intolerance, Pancreas
Keywords: Sodium-glucose transporter 2 inhibitor
MeSH Terms: conditions — Diabetes Mellitus; Platelet Glycoprotein IV Deficiency | interventions — empagliflozin; Sodium-Glucose Transporter 2 Inhibitors; Hypoglycemic Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (Active Comparator): up-titration of standard medication including monotherapy or combination of Metformin, Sulfonylurea, DPP4 inhibitor
  Interventions: Drug: Hypoglycemics Oral
- Study group (Experimental): addition of empagliflozin 10mg qd on standard oral antihyperglycemic agents
  Interventions: Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — addition of empagliflozin 10 MG
  Other Names: SGLT2 inhibitor
  Arms: Study group
Drug: Hypoglycemics Oral — dose escalation of hypoglycemics oral
  Other Names: Oral antidiabetic medication escalation
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate changes of body composition induced by Sodium-glucose cotransporter-2 (SGLT2) inhibitor and its metabolic consequence in Korean type 2 diabetes (T2D).

DETAILED DESCRIPTION:
Sodium-glucose cotransporter-2 (SGLT2) inhibitor increases urinary excretion of glucose, promoting glycemic control and weight loss. However, it is unclear whether weight loss is attributed to decrease in fat components and associated with favorable changes in metabolic profile. The purpose of this study is to evaluate changes of body composition induced by SGLT2 inhibitor and its metabolic consequence in Korean type 2 diabetes (T2D).

ELIGIBILITY:
Inclusion Criteria:

Patients with type 2 diabetes Age: 20-79 years BMI ≥ 20 kg/m2 eGFR ≥ 45

Exclusion Criteria:

Patients with type 1 diabetes Secondary diabetes due to Cushing diseases, acromegaly Insulin user BMI < 20 kg/m2 eGFR < 45 Malignancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 6 months
  glycemic control

SECONDARY OUTCOMES:
Biochemical parameters | 6 months
  Ketone body concentration
Body weight | 6 months
  Weight change
Body fat | 6 months
  fat change
Systolic and diastolic blood pressures | 6 months
  blood pressure change
Lipid profile | 6 months
  Triglyceride
Insulin resistance | 6 months
  HOMA-IR

CONTACTS AND LOCATIONS:
Overall Officials: Soo N Lim, MD, PHD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided